CLINICAL TRIAL: NCT03817463
Title: Multi-country Non-interventional Study on the Effectiveness of Empagliflozin in Adult Patients With Type 2 Diabetes in Europe and Asia.
Brief Title: A Study to Observe the Effectiveness of Empagliflozin, Other SGLT-2 Inhibitors, or DPP-4 Inhibitors in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0195
Record Dates: First submitted 2019-01-24; First posted 2019-01-25 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Sodium-Glucose Transporter 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New users of SGLT-2i: Patients with type 2 diabetes mellitus (T2DM), who were new users of any sodium-glucose cotransporter-2 inhibitors (SGLT-2i) including empagliflozin.
  Interventions: Drug: Subjects treated with Empagliflozin or any Sodium-glucose cotransporter-2 (SGLT-2) inhibitor
- New users of DPP-4i: Patients with type 2 diabetes mellitus (T2DM), who were new users of dipeptidyl peptidase-4 inhibitors (DPP-4i).
  Interventions: Drug: Subjects treated with Dipeptidyl peptidase-4 (DPP-4) inhibitor

INTERVENTIONS:
Drug: Subjects treated with Empagliflozin or any Sodium-glucose cotransporter-2 (SGLT-2) inhibitor — Empagliflozin or any Sodium-glucose cotransporter-2 (SGLT-2) inhibitor
  Groups: New users of SGLT-2i
Drug: Subjects treated with Dipeptidyl peptidase-4 (DPP-4) inhibitor — Dipeptidyl peptidase-4 (DPP-4) inhibitor
  Groups: New users of DPP-4i

SUMMARY:
Non-interventional, multi-country cohort study using existing data and including adults (≥18 years) with a diagnosis of Type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Dispensation or any other record of empagliflozin, any SGLT-2 inhibitor, or any DPP-4 inhibitor use during the study period
* No dispensation or any other record of any other SGLT-2 inhibitor or DPP-4 inhibitor use during the preceding 12 months including at index date
* Having a diagnosis of T2DM before the index date, based on ICD-10 codes or other available data

Exclusion Criteria:

* Aged <18 years on the first dispensation date or date of the first record of empagliflozin, any SGLT-2 inhibitor or any DPP-4 inhibitor use
* Type 1 diabetes mellitus
* Secondary diabetes
* Gestational diabetes
* Having a diagnosis of ESRD during the 12 months before the index date
* <12 months of available data before the index date, and/or no complete history of drug dispensations/other records of the drug use during this period
* Missing or ambiguous data on age or sex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a non-interventional, multi-country cohort study using existing data and including adults (≥18 years) with a diagnosis of T2DM. All data will be obtained from electronically recorded longitudinal secondary data sources, separately in each included country. In each country, patients initiating treatment with empagliflozin or any other SGLT-2 inhibitor will be compared with PS-matched patients initiating treatment with any DPP-4inhibitor.
Sampling Method: Probability Sample
Enrollment: 327624 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly G Brodovicz, (203) 448-1937, Study Chair — kimberly.brodovicz@boehringer-ingelheim.com
Locations (13):
- Steno Diabetes Center Copenhagen, Department of Clinical Epidemiology, Gentofte Municipality, Denmark
- Helsinki University Hospital, Helsinki, Finland
- University of Ulm, Institute for Epidemiology and medical biometry, Ulm, Germany
- Maccabi Healthcare Services, Tel Aviv, Israel
- Gifu University, Gifu, Japan
- Norway (2):
  - Oslo University Hospital, Department of Clinical Lipidology, Oslo
  - Oslo University Hospital, Department of Cardiology, Oslo
- Ajou University Hospital, Suwon, South Korea
- Instituto de Investigación Sanitaria INCLIVA, Valencia, Spain
- Sweden (2):
  - TFS Trial Form Support International AB, Lund
  - Quantify Research AB, Stockholm
- Taiwan Society for Pharmacoeconomics and Outcome Research (TaSPOR), Taipei, Taiwan
- Leicester Real World Evidence Unit, Leicester general Hospital, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Nystrom T, Toresson Grip E, Gunnarsson J, Casajust P, Karlsdotter K, Skogsberg J, Ustyugova A; EMPRISE Study Group. Empagliflozin reduces cardiorenal events, healthcare resource use and mortality in Sweden compared to dipeptidyl peptidase-4 inhibitors: Real world evidence from the Nordic EMPRISE study. Diabetes Obes Metab. 2023 Jan;25(1):261-271. doi: 10.1111/dom.14870. Epub 2022 Oct 10. PMID 36097728
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional, multi-country study to compare the effectiveness and safety of empagliflozin in adult patients with type 2 diabetes. The study used secondary data sources from eleven countries, identifying new users of empagliflozin, any SGLT-2 inhibitor or any DPP4-inhibitor from May 2014 or November 2012 until December 2019.
Pre-assignment Details: All subjects who strictly met all inclusion and none of the exclusion criteria where included in the study.
Groups:
- SGLT-2i (Incl. Empa) (Matched to DPP-4i): Patients with type 2 diabetes mellitus (T2DM), who were new users of any sodium-glucose cotransporter-2 inhibitors (SGLT-2i), including (incl.) new users of empagliflozin (empa). The study used secondary data sources from 11 countries (Denmark, Finland, Germany, Israel, Japan, Norway, South Korea, Spain, Sweden, Taiwan and the United Kingdom (UK CPRD, UK THIN) to identify new users of any SGLT-2i between November 2012 and December 2019. New user of any SGLT-2i were matched to new users of DPP-4i using a 1:1 propensity score (PS)-matching approach.
- DPP-4i (Matched to SGLT-2i): Patients with type 2 diabetes mellitus (T2DM), who were new users of dipeptidyl peptidase-4 inhibitors (DPP-4i). The study used secondary data sources from 11 countries (Denmark, Finland, Germany, Israel, Japan, Norway, South Korea, Spain, Sweden, Taiwan and the United Kingdom (UK CPRD, UK THIN) to identify new users of DPP-4i between November 2012 and December 2019. New users of DPP-4i where matched to new users of any SGLT-2i using a 1:1 propensity score (PS)-matching approach.
Period: Overall Study
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i)
Started | 163812 | 163812
Completed | 163812 | 163812
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients included in the study, who were either new user of any SGLT-2i (incl. empagliflozin) or DPP-4i.
Groups:
- Total: Total of all reporting groups
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Total
Number analyzed (Participants) | 163812 | 163812 | 327624
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.02 (12.49) | 59.55 (12.49) | 59.56 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70990 | 71002 | 141992
  Male | 92822 | 92810 | 185632
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hospitalization for Heart Failure (HHF), Broad + Specific Definition
Description: Number of participants with Hospitalization for Heart Failure (HHF), using broad + specific HHF definition.
  HHF - broad defined as any diagnosis associated with healthcare encounters, including hospitalizations and specialist outpatient and primary care encounters, or dispensation or any other record of the high-ceiling diuretics (loop diuretics).
  HHF - specific defined as a primary diagnosis associated with hospital admission.
  For HHF - broad + specific, HHF-specific definition was used unless only broad definition were available. However, for Japan South Korea and Taiwan, both definitions were available, but broad definition was used.
Time Frame: From index date until end of follow-up, up to 67 months for matched cohort of empagliflozin/DPP-4i. Up to 86 months for matched cohort of SGLT-2i/DPP-4i
Population: All patients included in the study, who were either new user of any SGLT-2i (incl. empagliflozin) or DPP-4i. Results are reported by 1:1 PS-matched cohorts of SGLT-2i/DPP-4i and empagliflozin/DPP-4i. Arms are not mutually exclusive.
Measure: Count of Participants; unit: Participants
Groups:
- Empagliflozin (Matched to DPP-4i): Patients with type 2 diabetes mellitus (T2DM), who were new users of empagliflozin between May 2014 and December 2019, identified from secondary data sources from 11 countries. New users of empagliflozin were matched to new users of DPP-4i using a propensity score (PS)-matching approach.
- DPP-4i (Matched to Empagliflozin): Patients with type 2 diabetes mellitus (T2DM), who were new users of dipeptidyl peptidase-4 inhibitors (DPP-4i) between May 2014 and December 2019, identified from secondary data sources from 11 countries. DPP-4 users were matched to new users of empagliflozin, using a 1:1 propensity score matching approach.
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 163812 | 163812 | 85244 | 85244
Participants | 1395 | 2043 | 765 | 1083
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); HHF-(broad+specific); Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.70, 95% CI 2-sided [0.60 to 0.83]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); HHF-(broad + specific); Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.66, 95% CI 2-sided [0.57 to 0.78]

2. Primary Outcome: Number of Participants With Hospitalization for Heart Failure (HHF), Broad Definition
Description: Reported is the number of participants with hospitalization for heart failure (HHF), using broad definition of HHF.
  HHF - broad is defined as any diagnosis associated with healthcare encounters, including hospitalizations and specialist outpatient and primary care encounters, or dispensation or any other record of the high-ceiling diuretics (loop diuretics).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 163812 | 163812 | 85244 | 85244
Participants | 964 | 1260 | 514 | 641
Statistical Analysis 1: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); HHF-broad; Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Ajusted hazard ratio = 0.75, 95% CI 2-sided [0.69 to 0.81]
Statistical Analysis 2: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); HHF-broad; Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Ajusted hazard ratio = 0.78, 95% CI 2-sided [0.69 to 0.88]

3. Primary Outcome: Number of Participants With Hospitalization for Heart Failure (HHF), Specific Definition
Description: Reported is the number of participants with hospitalization for heart failure, using specific definition for HHF.
  HHF - specific defined as a primary diagnosis associated with hospital admission.
Time Frame: as for outcome 1
Population: Patients, who were either new user of any SGLT-2i (incl. empagliflozin) or DPP-4i. Results are reported by 1:1 PS-matched cohorts of SGLT-2i/DPP-4i and empagliflozin/DPP-4i. Arms are not mutually exclusive. Country-level results are reported and only include countries with non-missing data or a sufficient number of events to satisfy local patient privacy regulations.
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 144306 | 144306 | 68087 | 68087
Participants
  Denmark: number analyzed (Participants) | 15459 | 15459 | 9765 | 9765
  Denmark | 273 | 345 | 178 | 195
  Finnland: number analyzed (Participants) | 16917 | 16917 | 11801 | 11801
  Finnland | 80 | 190 | 53 | 128
  Germany: number analyzed (Participants) | 1687 | 1687 | 839 | 839
  Germany | 33 | 76 | 18 | 35
  Israel: number analyzed (Participants) | 5064 | 5064 | 3913 | 3913
  Israel | 27 | 28 | 25 | 27
  Japan: number analyzed (Participants) | 12985 | 12985 | 5592 | 5592
  Japan | 105 | 114 | 59 | 65
  South Korea: number analyzed (Participants) | 22852 | 22852 | 0 | 0
  South Korea | 12 | 19 |  |
  Norway: number analyzed (Participants) | 12510 | 12510 | 6344 | 6344
  Norway | 49 | 124 | 23 | 63
  Sweden: number analyzed (Participants) | 22436 | 22436 | 15785 | 15785
  Sweden | 106 | 200 | 59 | 127
  Taiwan: number analyzed (Participants) | 34396 | 34396 | 14048 | 14048
  Taiwan | 60 | 86 | 29 | 38
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); HHF-specific. Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.68, 95% CI 2-sided [0.56 to 0.83]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); HHF-specific. Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.64, 95% CI 2-sided [0.51 to 0.81]

4. Primary Outcome: Number of Participants With All-cause Mortality (ACM)
Description: Number of participants with all-cause mortality (ACM).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 163812 | 163812 | 85244 | 85244
Participants | 1371 | 2524 | 572 | 1177
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.55, 95% CI 2-sided [0.48 to 0.63]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.59, 95% CI 2-sided [0.54 to 0.65]

5. Primary Outcome: Number of Participants With Composite Outcome, Including Hospitalization for Heart Failure (HHF) and All Cause Mortality (ACM)
Description: Number of participants with composite outcome, including hospitalization for heart failure (HHF) and all cause mortality (ACM).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 163812 | 163812 | 85244 | 85244
Participants | 2413 | 3749 | 1239 | 2063
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Test type: Other; p < 0.05, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.65, 95% CI 2-sided [0.56 to 0.76]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.66, 95% CI 2-sided [0.61 to 0.72]

6. Primary Outcome: Number of Participants With Composite Outcome, Including Myocardial Infraction (MI), Stroke and All Cause Mortality (ACM)
Description: Number of participants with composite outcome, including myocardial infraction (MI), stroke and all cause mortality (ACM).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 163812 | 163812 | 85244 | 85244
Participants | 2548 | 3758 | 1236 | 1950
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.72, 95% CI 2-sided [0.64 to 0.82]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.72, 95% CI 2-sided [0.66 to 0.78]

7. Primary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: Number of participants with myocardial infarction (MI).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Empagliflozin (Matched to DPP-4i): PPatients with type 2 diabetes mellitus (T2DM), who were new users of empagliflozin between May 2014 and December 2019, identified from secondary data sources from 11 countries. New users of empagliflozin were matched to new users of DPP-4i using a propensity score (PS)-matching approach.
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 163812 | 163812 | 85244 | 85244
Participants | 701 | 863 | 364 | 414
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Test type: Other; p = 0.816, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 1.02, 95% CI 2-sided [0.88 to 1.18]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Test type: Other; p = 0.013, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.87, 95% CI 2-sided [0.78 to 0.97]

8. Primary Outcome: Number of Participants With Stroke
Description: Number of participants with stroke.
Time Frame: as for outcome 1
Population: All patients included in the study, who were either new user of any SGLT-2i (incl. empagliflozin) or DPP-4i. Results are reported by 1:1 PS-matched cohorts of SGLT-2i/DPP-4i and empagliflozin/DPP-4i. Arms are not mutually exclusive. Country-level results are reported and only include countries with non-missing data or a sufficient number of events to satisfy local patient privacy regulations.
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 163812 | 163812 | 84405 | 84405
Participants
  Denmark: number analyzed (Participants) | 15459 | 15459 | 9765 | 9765
  Denmark | 183 | 230 | 110 | 112
  Finland: number analyzed (Participants) | 16917 | 16917 | 11801 | 11801
  Finland | 38 | 54 | 24 | 40
  Germany: number analyzed (Participants) | 1687 | 1687 | 0 | 0
  Germany | 6 | 24 |  |
  Israel: number analyzed (Participants) | 5064 | 5064 | 3913 | 3913
  Israel | 20 | 21 | 15 | 17
  Japan: number analyzed (Participants) | 12985 | 12985 | 5592 | 5592
  Japan | 26 | 50 | 12 | 13
  South Korea: number analyzed (Participants) | 22852 | 22852 | 9072 | 9072
  South Korea | 107 | 187 | 43 | 68
  Norway: number analyzed (Participants) | 12510 | 12510 | 6344 | 6344
  Norway | 72 | 87 | 28 | 36
  Spain: number analyzed (Participants) | 12899 | 12899 | 5865 | 5865
  Spain | 49 | 53 | 15 | 27
  Sweden: number analyzed (Participants) | 22436 | 22436 | 15785 | 15785
  Sweden | 120 | 134 | 53 | 102
  Taiwan: number analyzed (Participants) | 34396 | 34396 | 14048 | 14048
  Taiwan | 118 | 104 | 53 | 53
  UK Clinical Practice Research Datalink (CPRD): number analyzed (Participants) | 2718 | 2718 | 922 | 922
  UK Clinical Practice Research Datalink (CPRD) | 42 | 39 | 12 | 12
  UK the Health Improvement Network databases (THIN): number analyzed (Participants) | 3889 | 3889 | 1298 | 1298
  UK the Health Improvement Network databases (THIN) | 17 | 0 | 7 | 6
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p < 0.011, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.82, 95% CI 2-sided [0.71 to 0.96]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p = 0.064, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.84, 95% CI 2-sided [0.69 to 1.01]

9. Secondary Outcome: Number of Participants With Cardiovascular Mortality (CM)
Description: Number of participants with cardiovascular mortality (CM).
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 86259 | 86259 | 47978 | 47978
Participants
  Finland: number analyzed (Participants) | 16917 | 16917 | 11801 | 11801
  Finland | 67 | 161 | 35 | 107
  Norway: number analyzed (Participants) | 12510 | 12510 | 6344 | 6344
  Norway | 44 | 73 | 17 | 32
  Sweden: number analyzed (Participants) | 22436 | 22436 | 15785 | 15785
  Sweden | 56 | 109 | 24 | 80
  Taiwan: number analyzed (Participants) | 34396 | 34396 | 14048 | 14048
  Taiwan | 53 | 76 | 28 | 29
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.59, 95% CI 2-sided [0.42 to 0.84]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.60, 95% CI 2-sided [0.49 to 0.72]

10. Secondary Outcome: Number of Participants With Composite Outcome Including Hospitalization for Heart Failure (HHF) and Cardiovascular (CV) Mortality
Description: Number of participants with composite outcome including hospitalization for heart failure (HHF) and cardiovascular (CV) mortality.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 163812 | 163812 | 85244 | 85244
Participants | 397 | 806 | 205 | 505
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.54, 95% CI 2-sided [0.46 to 0.64]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.56, 95% CI 2-sided [0.47 to 0.66]

11. Secondary Outcome: Number of Participants With 3-point Major Adverse Cardiovascular (CV) Events (MACE), Defined as a Composite Outcome Including Myocardial Infarction (MI), Stroke and Cardiovascular (CV) Mortality
Description: Number of participants with 3-point major adverse cardiovascular (CV) events (MACE), defined as a composite outcome including myocardial infarction (MI), stroke and cardiovascular (CV) mortality.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 163812 | 163812 | 85244 | 85244
Participants | 843 | 1009 | 393 | 516
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Test type: Other; p = 0.545, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.95, 95% CI 2-sided [0.81 to 1.11]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Test type: Other; p = 0.036, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.91, 95% CI 2-sided [0.83 to 0.99]

12. Secondary Outcome: Number of Participants With Coronary Revascularization Procedure
Description: Number of participants with coronary revascularization procedure.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Empagliflozin (Matched to DPP-4i): Patients with type 2 diabetes mellitus (T2DM), who were new users of empagliflozin between May 2014 and December 2019, in all countries included in this study. Empagliflozin users were matched to incident users of (dipeptidyl peptidase-4 inhibitors) DPP-4i using a 1:1 propensity score matching approach.
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 159923 | 159923 | 77242 | 77242
Participants
  Denmark: number analyzed (Participants) | 15459 | 15459 | 9765 | 9765
  Denmark | 173 | 184 | 117 | 109
  Finland: number analyzed (Participants) | 16917 | 16917 | 11801 | 11801
  Finland | 26 | 19 | 12 | 15
  Germany: number analyzed (Participants) | 1687 | 1687 | 0 | 0
  Germany | 9 | 20 |  |
  Israel: number analyzed (Participants) | 5064 | 5064 | 3913 | 3913
  Israel | 124 | 103 | 111 | 89
  Japan: number analyzed (Participants) | 12985 | 12985 | 5592 | 5592
  Japan | 268 | 383 | 158 | 206
  South Korea: number analyzed (Participants) | 22852 | 22852 | 9072 | 9072
  South Korea | 66 | 97 | 23 | 33
  Norway: number analyzed (Participants) | 12510 | 12510 | 6344 | 6344
  Norway | 58 | 64 | 10 | 11
  Spain: number analyzed (Participants) | 12899 | 12899 | 0 | 0
  Spain | 0 | 7 |  |
  Sweden: number analyzed (Participants) | 22436 | 22436 | 15785 | 15785
  Sweden | 212 | 263 | 115 | 153
  Taiwan: number analyzed (Participants) | 34396 | 34396 | 14048 | 14048
  Taiwan | 296 | 280 | 140 | 152
  UK Clinical Practice Research Datalink (CPRD): number analyzed (Participants) | 2718 | 2718 | 922 | 922
  UK Clinical Practice Research Datalink (CPRD) | 61 | 73 | 13 | 18
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p = 0.353, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.93, 95% CI 2-sided [0.79 to 1.09]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p = 0.197, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.90, 95% CI 2-sided [0.78 to 1.05]

13. Secondary Outcome: Number of Participants With End-stage Renal Disease (ESRD)
Description: Number of participants with end-stage renal disease (ESRD).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 119397 | 119397 | 56143 | 56143
Participants
  Denmark: number analyzed (Participants) | 15459 | 15459 | 9765 | 9765
  Denmark | 65 | 116 | 34 | 56
  Finland: number analyzed (Participants) | 16917 | 16917 | 11801 | 11801
  Finland | 14 | 43 | 8 | 25
  Japan: number analyzed (Participants) | 12985 | 12985 | 5592 | 5592
  Japan | 8 | 37 | 6 | 17
  South Korea: number analyzed (Participants) | 22852 | 22852 | 9072 | 9072
  South Korea | 0 | 21 | 0 | 9
  Spain: number analyzed (Participants) | 12899 | 12899 | 5865 | 5865
  Spain | 0 | 9 | 0 | 5
  Taiwan: number analyzed (Participants) | 34396 | 34396 | 14048 | 14048
  Taiwan | 38 | 131 | 21 | 52
  UK Health Improvement Network databases (THIN): number analyzed (Participants) | 3889 | 3889 | 0 | 0
  UK Health Improvement Network databases (THIN) | 0 | 5 |  |
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.43, 95% CI 2-sided [0.30 to 0.63]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.27, 95% CI 2-sided [0.16 to 0.44]

14. Secondary Outcome: Number of Participants With Estimated Glomerular Filtration Rate (eGFR) Decline
Description: Number of participants with estimated glomerular filtration rate (eGFR) decline.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 163812 | 163812 | 85244 | 85244
Participants | 1569 | 1908 | 914 | 1043
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Test type: Other; p = 0.535, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 1.05, 95% CI 2-sided [0.89 to 1.25]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Test type: Other; p = 0.850, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.98, 95% CI 2-sided [0.84 to 1.15]

15. Secondary Outcome: Number of Participants With Progression From Normoalbuminuria to Micro- or Macroalbuminuria
Description: Number of participants with progression from normoalbuminuria to micro- or macroalbuminuria.
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 14080 | 14080 | 8509 | 8509
Participants
  Germany: number analyzed (Participants) | 1269 | 1269 | 614 | 614
  Germany | 260 | 158 | 121 | 79
  Israel: number analyzed (Participants) | 2973 | 2973 | 2318 | 2318
  Israel | 215 | 213 | 165 | 149
  Sweden: number analyzed (Participants) | 6696 | 6696 | 4926 | 4926
  Sweden | 297 | 401 | 149 | 257
  UK Clinical Practice Research Datalink (CPRD): number analyzed (Participants) | 1084 | 1084 | 344 | 344
  UK Clinical Practice Research Datalink (CPRD) | 55 | 79 | 19 | 18
  UK Health Improvement Network databases (THIN): number analyzed (Participants) | 2058 | 2058 | 0 | 0
  UK Health Improvement Network databases (THIN) | 15 | 24 |  |
  Finland: number analyzed (Participants) | 0 | 0 | 307 | 307
  Finland |  |  | 6 | 6
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p = 0.828, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 1.03, 95% CI 2-sided [0.81 to 1.31]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p = 0.944, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 1.01, 95% CI 2-sided [0.72 to 1.42]

16. Secondary Outcome: Number of Participants With Composite Outcome Including eGFR Decline and Progression to Micro- or Macroalbuminuria
Description: Number of participants with composite outcome including Estimated glomerular filtration rate (eGFR) decline and progression to micro- or macroalbuminuria.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i) | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 163812 | 163812 | 85244 | 85244
Participants | 2456 | 3652 | 1324 | 1710
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Test type: Other; p = 0.642, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.94, 95% CI 2-sided [0.73 to 1.22]
Statistical Analysis 2: Comparison: SGLT-2i (Incl. Empa) (Matched to DPP-4i) vs DPP-4i (Matched to SGLT-2i); Test type: Other; p = 0.417, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.89, 95% CI 2-sided [0.66 to 1.19]

17. Secondary Outcome: Number of Participants With Bone Fracture
Description: Number of participants with bone fracture. Data for this endpoint was only collected and analyzed for the matched cohort of empagliflozin/DPP-4i.
Time Frame: From index date until end of follow-up, up to 67 months.
Population: Only patients in the study, who were included in the 1:1 propensity-score matched cohort of empagliflozin/DPP-4i. Country-level results are reported and only include countries with non-missing data or a sufficient number of events to satisfy local patient privacy regulations.
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 82185 | 82185
Participants
  Denmark: number analyzed (Participants) | 9765 | 9765
  Denmark | 91 | 88
  Finland: number analyzed (Participants) | 11801 | 11801
  Finland | 40 | 59
  Israel: number analyzed (Participants) | 3913 | 3913
  Israel | 10 | 6
  Japan: number analyzed (Participants) | 5592 | 5592
  Japan | 6 | 11
  South Korea: number analyzed (Participants) | 9072 | 9072
  South Korea | 41 | 50
  Norway: number analyzed (Participants) | 6344 | 6344
  Norway | 23 | 45
  Spain: number analyzed (Participants) | 5865 | 5865
  Spain | 19 | 20
  Sweden: number analyzed (Participants) | 15785 | 15785
  Sweden | 66 | 98
  Taiwan: number analyzed (Participants) | 14048 | 14048
  Taiwan | 47 | 50
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p = 0.091, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.89, 95% CI 2-sided [0.77 to 1.02]

18. Secondary Outcome: Number of Participants With Diabetic Ketoacidosis
Description: Number of participants with diabetic ketoacidosis. Data for this endpoint was only collected and analyzed for the matched cohort of empagliflozin/DPP-4i
Time Frame: From index date until end of follow-up, up to 67 months.
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Groups:
- DPP-4i (Matched to Empagliflozin): Patients with type 2 diabetes mellitus (T2DM), who were new users of dipeptidyl peptidase-4 inhibitors (DPP-4i) between May 2014 and December 2019, identified from secondary data sources from eleven countries. DPP-4 users were matched to new users of empagliflozin, using a 1:1 propensity score matching approach.
Arm/Group | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 40896 | 40896
Participants
  Denmark: number analyzed (Participants) | 9765 | 9765
  Denmark | 16 | 6
  Sweden: number analyzed (Participants) | 15785 | 15785
  Sweden | 16 | 11
  Taiwan: number analyzed (Participants) | 14048 | 14048
  Taiwan | 19 | 9
  UK Health Improvement Network databases (THIN): number analyzed (Participants) | 1298 | 1298
  UK Health Improvement Network databases (THIN) | 5 | 0
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 1.97, 95% CI 2-sided [1.28 to 3.03]

19. Secondary Outcome: Number of Participants With Severe Hypoglycemia
Description: Number of participants with severe hypoglycemia. Data for this endpoint was only collected and analyzed for the matched cohort of empagliflozin/DPP-4i.
Time Frame: From index date until end of follow-up, up to 67 months.
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 73308 | 73308
Participants
  Denmark: number analyzed (Participants) | 9765 | 9765
  Denmark | 29 | 23
  Finland: number analyzed (Participants) | 11801 | 11801
  Finland | 11 | 13
  Germany: number analyzed (Participants) | 839 | 839
  Germany | 16 | 7
  Israel: number analyzed (Participants) | 3913 | 3913
  Israel | 24 | 22
  South Korea: number analyzed (Participants) | 9072 | 9072
  South Korea | 12 | 18
  Spain: number analyzed (Participants) | 5865 | 5865
  Spain | 14 | 14
  Sweden: number analyzed (Participants) | 15785 | 15785
  Sweden | 11 | 17
  Taiwan: number analyzed (Participants) | 14048 | 14048
  Taiwan | 229 | 294
  UK Clinical Practice Research Datalink (CPRD): number analyzed (Participants) | 922 | 922
  UK Clinical Practice Research Datalink (CPRD) | 0 | 0
  UK Health Improvement Network databases (THIN): number analyzed (Participants) | 1298 | 1298
  UK Health Improvement Network databases (THIN) | 5 | 9
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p = 0.654, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.95, 95% CI 2-sided [0.75 to 1.20]

20. Secondary Outcome: Number of Participants With Lower-limb Amputation
Description: Number of participants with lower-limb amputation. Data for this endpoint was only collected and analyzed for the matched cohort of empagliflozin/DPP-4i.
Time Frame: From index date until end of follow-up, up to 67 months.
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 40437 | 40437
Participants
  Denmark: number analyzed (Participants) | 9765 | 9765
  Denmark | 9 | 8
  Germany: number analyzed (Participants) | 839 | 839
  Germany | 12 | 16
  Sweden: number analyzed (Participants) | 15785 | 15785
  Sweden | 5 | 8
  Taiwan: number analyzed (Participants) | 14048 | 14048
  Taiwan | 6 | 11
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p = 0.233, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.78, 95% CI 2-sided [0.52 to 1.17]

21. Secondary Outcome: Number of Participants With Acute Kidney Injury Requiring Dialysis
Description: Number of participants with acute kidney injury requiring dialysis. Data for this endpoint was only collected and analyzed for the matched cohort of empagliflozin/DPP-4i.
Time Frame: From index date until end of follow-up, up to 67 months.
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Empagliflozin (Matched to DPP-4i) | DPP-4i (Matched to Empagliflozin)
Number analyzed (Participants) | 29678 | 29678
Participants
  Denmark: number analyzed (Participants) | 9765 | 9765
  Denmark | 33 | 40
  Spain: number analyzed (Participants) | 5865 | 5865
  Spain | 21 | 46
  Taiwan: number analyzed (Participants) | 14048 | 14048
  Taiwan | 60 | 100
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4i) vs DPP-4i (Matched to Empagliflozin); Hazards ratios reported include data from all countries with non-missing values; Test type: Other; p < 0.005, Cox proportional hazard model; Cox proportional hazard model adjusted for unbalanced propensity score (PS)-variables at baseline; Adjusted Hazard Ratio = 0.56, 95% CI 2-sided [0.38 to 0.82]

22. Secondary Outcome: Healthcare Resource Utilization (HCRU): Number of Any Medical Visit
Description: HCRU data were collected from seven of the 11 participating countries including Finland, Japan, South Korea, Norway, Spain, Sweden, and Taiwan. Outcomes captured as HCRU include emergency room visits, first inpatient stay, all-cause hospital admissions and outpatient healthcare visits.
  HCRU outcomes were investigated for the matched cohort of empagliflozin/DPP-4 only. Due to possibly huge differences in healthcare systems and local practices, HCRU outcomes were presented descriptively by country as per prespecified analysis plan.
  For arms with 0 patients analyzed, no data was collected for the specific outcome in this country.
Time Frame: From index date until end of follow-up, up to 67 months.
Population: Only patients in the study, who were included in the matched cohort of empagliflozin/DPP-4i from the following seven countries: Finland, Japan, South Korea, Norway, Spain, Sweden or Taiwan. HCRU outcomes are presented descriptively by country as per prespecified analysis plan. For arms with 0 patients analyzed, no data was collected for the specific outcome in this country.
Measure: Number; unit: Visit
Groups:
- Empagliflozin (Matched to DPP-4) - Finland: Patients with type 2 diabetes mellitus (T2DM), who were new users of empagliflozin between May 2014 and December 2019. Empagliflozin users were matched to incident users of (dipeptidyl peptidase-4) DPP-4 using a 1:1 propensity score matching approach. Only finish patients are included in this group.
- DPP-4 (Matched to Empagliflozin) - Finland: Patients with type 2 diabetes mellitus (T2DM), who were new users of dipeptidyl peptidase-4 (DPP-4) between May 2014 and December 2019, in all countries included in this study. DPP-4 users were matched to incident users of empagliflozin, using a 1:1 propensity score matching approach.
  Only finish patients are included in this arm
- Empagliflozin (Matched to DPP-4) - Japan: Patients with type 2 diabetes mellitus (T2DM), who were new users of empagliflozin between May 2014 and December 2019, in all countries included in this study. Empagliflozin users were matched to incident users of (dipeptidyl peptidase-4) DPP-4 using a 1:1 propensity score matching approach.
  Only japanese patients are included in this arm.
- DPP-4 (Matched to Empagliflozin) - Japan: Patients with type 2 diabetes mellitus (T2DM), who were new users of dipeptidyl peptidase-4 (DPP-4) between May 2014 and December 2019, in all countries included in this study. DPP-4 users were matched to incident users of empagliflozin, using a 1:1 propensity score matching approach.
  Only japanese patients are included in this arm.
- Empagliflozin (Matched to DPP-4) - South Korea: Patients with type 2 diabetes mellitus (T2DM), who were new users of empagliflozin between May 2014 and December 2019, in all countries included in this study. Empagliflozin users were matched to incident users of (dipeptidyl peptidase-4) DPP-4 using a 1:1 propensity score matching approach.
  Only south-korean patients are included in this arm.
- DPP-4 (Matched to Empagliflozin) - South Korea: Patients with type 2 diabetes mellitus (T2DM), who were new users of dipeptidyl peptidase-4 (DPP-4) between May 2014 and December 2019, in all countries included in this study. DPP-4 users were matched to incident users of empagliflozin, using a 1:1 propensity score matching approach.
  Only south-korean patients are included in this arm.
- Empagliflozin (Matched to DPP-4) - Norway: Patients with type 2 diabetes mellitus (T2DM), who were new users of empagliflozin between May 2014 and December 2019, in all countries included in this study. Empagliflozin users were matched to incident users of (dipeptidyl peptidase-4) DPP-4 using a 1:1 propensity score matching approach.
  Only norwegian patients are included in this arm.
- DPP-4 (Matched to Empagliflozin) - Norway: Patients with type 2 diabetes mellitus (T2DM), who were new users of dipeptidyl peptidase-4 (DPP-4) between May 2014 and December 2019, in all countries included in this study. DPP-4 users were matched to incident users of empagliflozin, using a 1:1 propensity score matching approach.
  Only norwegian patients are included in this arm.
- Empagliflozin (Matched to DPP-4) - Spain: Patients with type 2 diabetes mellitus (T2DM), who were new users of empagliflozin between May 2014 and December 2019, in all countries included in this study. Empagliflozin users were matched to incident users of (dipeptidyl peptidase-4) DPP-4 using a 1:1 propensity score matching approach.
  Only spanish patients are included in this arm.
- DPP-4 (Matched to Empagliflozin) - Spain: Patients with type 2 diabetes mellitus (T2DM), who were new users of dipeptidyl peptidase-4 (DPP-4) between May 2014 and December 2019, in all countries included in this study. DPP-4 users were matched to incident users of empagliflozin, using a 1:1 propensity score matching approach.
  Only spanish patients are included in this arm.
- Empagliflozin (Matched to DPP-4) - Sweden: Patients with type 2 diabetes mellitus (T2DM), who were new users of empagliflozin between May 2014 and December 2019, in all countries included in this study. Empagliflozin users were matched to incident users of (dipeptidyl peptidase-4) DPP-4 using a 1:1 propensity score matching approach.
  Only swedish patients are included in this arm.
- DPP-4 (Matched to Empagliflozin) - Sweden: Patients with type 2 diabetes mellitus (T2DM), who were new users of dipeptidyl peptidase-4 (DPP-4) between May 2014 and December 2019, in all countries included in this study. DPP-4 users were matched to incident users of empagliflozin, using a 1:1 propensity score matching approach.
  Only swedish patients are included in this arm.
- Empagliflozin (Matched to DPP-4) - Taiwan: Patients with type 2 diabetes mellitus (T2DM), who were new users of empagliflozin between May 2014 and December 2019, in all countries included in this study. Empagliflozin users were matched to incident users of (dipeptidyl peptidase-4) DPP-4 using a 1:1 propensity score matching approach.
  Only taiwanese patients are included in this arm.
- DPP-4 (Matched to Empagliflozin) - Taiwan: Patients with type 2 diabetes mellitus (T2DM), who were new users of dipeptidyl peptidase-4 (DPP-4) between May 2014 and December 2019, in all countries included in this study. DPP-4 users were matched to incident users of empagliflozin, using a 1:1 propensity score matching approach.
  Only taiwanese patients are included in this arm.
Arm/Group | Empagliflozin (Matched to DPP-4) - Finland | DPP-4 (Matched to Empagliflozin) - Finland | Empagliflozin (Matched to DPP-4) - Japan | DPP-4 (Matched to Empagliflozin) - Japan | Empagliflozin (Matched to DPP-4) - South Korea | DPP-4 (Matched to Empagliflozin) - South Korea | Empagliflozin (Matched to DPP-4) - Norway | DPP-4 (Matched to Empagliflozin) - Norway | Empagliflozin (Matched to DPP-4) - Spain | DPP-4 (Matched to Empagliflozin) - Spain | Empagliflozin (Matched to DPP-4) - Sweden | DPP-4 (Matched to Empagliflozin) - Sweden | Empagliflozin (Matched to DPP-4) - Taiwan | DPP-4 (Matched to Empagliflozin) - Taiwan
Number analyzed (Participants) | 11801 | 11801 | 5592 | 5592 | 9072 | 9072 | 6344 | 6344 | 5865 | 5865 | 15785 | 15785 | 14048 | 14048
Visit
  Emergency room visis: number analyzed (Participants) | 11801 | 11801 | 5592 | 5592 | 9072 | 9072 | 0 | 0 | 5865 | 5865 | 15785 | 15785 | 14048 | 14048
  Emergency room visis | 1187 | 2138 | 42 | 43 | 767 | 847 |  |  | 178 | 228 | 1000 | 1613 | 2459 | 2834
  First inpatient stay | 1472 | 2294 | 582 | 704 | 1008 | 1266 | 885 | 1169 | 303 | 365 | 1401 | 2230 | 1192 | 1430
  All-caused hospital admissions | 2607 | 5147 | 747 | 1000 | 1499 | 2137 | 2191 | 3368 | 441 | 594 | 2413 | 4310 | 1620 | 2029
  Outpatient healthcare visits | 22232 | 38106 | 27521 | 26095 | 117437 | 121503 | 19543 | 25541 | 6191 | 6478 | 17590 | 27888 | 186380 | 191095
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4) - Finland vs DPP-4 (Matched to Empagliflozin) - Finland; Emergency room visits - Finland; Test type: Other; Rate Ratio = 0.74, 95% CI 2-sided [0.69 to 0.80] — Poisson regression model was used
Statistical Analysis 2: Comparison: Empagliflozin (Matched to DPP-4) - Japan vs DPP-4 (Matched to Empagliflozin) - Japan; Emergency room visits - Japan; Test type: Other; Rate Ratio = 0.90, 95% CI 2-sided [0.59 to 1.38] — Poisson regression model was used
Statistical Analysis 3: Comparison: Empagliflozin (Matched to DPP-4) - South Korea vs DPP-4 (Matched to Empagliflozin) - South Korea; Emergency room visits - South Korea; Test type: Other; Rate Ratio = 0.91, 95% CI 2-sided [0.82 to 1.00] — Poisson regression model was used
Statistical Analysis 4: Comparison: Empagliflozin (Matched to DPP-4) - Spain vs DPP-4 (Matched to Empagliflozin) - Spain; Emergency room visit - Spain; Test type: Other; Rate Ratio = 0.72, 95% CI 2-sided [0.59 to 0.87] — Poisson regression model was used
Statistical Analysis 5: Comparison: Empagliflozin (Matched to DPP-4) - Sweden vs DPP-4 (Matched to Empagliflozin) - Sweden; Emergency room visit - Sweden; Test type: Other; Rate Ratio = 0.94, 95% CI 2-sided [0.87 to 1.01] — Poisson regression model was used
Statistical Analysis 6: Comparison: Empagliflozin (Matched to DPP-4) - Taiwan vs DPP-4 (Matched to Empagliflozin) - Taiwan; Emergency room visit - Taiwan; Test type: Other; Rate Ratio = 0.86, 95% CI 2-sided [0.80 to 0.93] — Poisson regression model was used
Statistical Analysis 7: Comparison: Empagliflozin (Matched to DPP-4) - Finland vs DPP-4 (Matched to Empagliflozin) - Finland; First impatient stay - Finland; Test type: Other; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.75 to 0.85] — HR and confidence interval were estimated using a cox proportional hazard model, comparing treatment groups and adjusting for unbalanced propensity score (PS)-variables
Statistical Analysis 8: Comparison: Empagliflozin (Matched to DPP-4) - Japan vs DPP-4 (Matched to Empagliflozin) - Japan; First impatient stay - Japan; Test type: Other; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.68 to 0.84] — [estimate comment as in outcome 22, analysis 7]
Statistical Analysis 9: Comparison: Empagliflozin (Matched to DPP-4) - South Korea vs DPP-4 (Matched to Empagliflozin) - South Korea; First impatient stay - South Korea; Test type: Other; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.69 to 0.82] — [estimate comment as in outcome 22, analysis 7]
Statistical Analysis 10: Comparison: Empagliflozin (Matched to DPP-4) - Norway vs DPP-4 (Matched to Empagliflozin) - Norway; First impatient stay - Norway; Test type: Other; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.78 to 0.94] — [estimate comment as in outcome 22, analysis 7]
Statistical Analysis 11: Comparison: Empagliflozin (Matched to DPP-4) - Spain vs DPP-4 (Matched to Empagliflozin) - Spain; First impatient stay - Spain; Test type: Other; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.66 to 0.89] — [estimate comment as in outcome 22, analysis 7]
Statistical Analysis 12: Comparison: Empagliflozin (Matched to DPP-4) - Sweden vs DPP-4 (Matched to Empagliflozin) - Sweden; First impatient stay - Sweden; Test type: Other; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.81 to 0.93] — [estimate comment as in outcome 22, analysis 7]
Statistical Analysis 13: Comparison: Empagliflozin (Matched to DPP-4) - Taiwan vs DPP-4 (Matched to Empagliflozin) - Taiwan; First impatient stay - Taiwan; Test type: Other; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.74 to 0.86] — [estimate comment as in outcome 22, analysis 7]
Statistical Analysis 14: Comparison: Empagliflozin (Matched to DPP-4) - Finland vs DPP-4 (Matched to Empagliflozin) - Finland; All-cause hospital admissions; Test type: Other; Rate Ratio = 0.68, 95% CI 2-sided [0.64 to 0.71] — Poisson regression model was used
Statistical Analysis 15: Comparison: Empagliflozin (Matched to DPP-4) - Japan vs DPP-4 (Matched to Empagliflozin) - Japan; For all-cause hospital admissions - Japan; Test type: Other; Rate Ratio = 0.69, 95% CI 2-sided [0.63 to 0.76] — Poisson regression model was used
Statistical Analysis 16: Comparison: Empagliflozin (Matched to DPP-4) - South Korea vs DPP-4 (Matched to Empagliflozin) - South Korea; All-cause hospital admissions - South Korea; Test type: Other; Rate Ratio = 0.70, 95% CI 2-sided [0.66 to 0.75] — Poisson regression model was used
Statistical Analysis 17: Comparison: Empagliflozin (Matched to DPP-4) - Norway vs DPP-4 (Matched to Empagliflozin) - Norway; All-cause hospital admissions - Norway; Test type: Other; Rate Ratio = 0.81, 95% CI 2-sided [0.77 to 0.85] — Poisson regression model was used
Statistical Analysis 18: Comparison: Empagliflozin (Matched to DPP-4) - Spain vs DPP-4 (Matched to Empagliflozin) - Spain; All-cause hospital admissions - Spain; Test type: Other; Rate Ratio = 0.68, 95% CI 2-sided [0.60 to 0.77] — Poisson regression model was used
Statistical Analysis 19: Comparison: Empagliflozin (Matched to DPP-4) - Sweden vs DPP-4 (Matched to Empagliflozin) - Sweden; All-cause hospital admissions - Sweden; Test type: Other; Rate Ratio = 0.85, 95% CI 2-sided [0.80 to 0.89] — Poisson regression model was used
Statistical Analysis 20: Comparison: Empagliflozin (Matched to DPP-4) - Taiwan vs DPP-4 (Matched to Empagliflozin) - Taiwan; All-cause hospital admissions - Taiwan; Test type: Other; Rate Ratio = 0.79, 95% CI 2-sided [0.72 to 0.87]
Statistical Analysis 21: Comparison: Empagliflozin (Matched to DPP-4) - Finland vs DPP-4 (Matched to Empagliflozin) - Finland; Outpatient healthcare visits - Finland; Test type: Other; Rate Ratio = 0.78, 95% CI 2-sided [0.77 to 0.79] — Poisson regression model was used
Statistical Analysis 22: Comparison: Empagliflozin (Matched to DPP-4) - Japan vs DPP-4 (Matched to Empagliflozin) - Japan; Outpatient healthcare visits - Japan; Test type: Other; Rate Ratio = 0.95, 95% CI 2-sided [0.94 to 0.97] — Poisson regression model was used
Statistical Analysis 23: Comparison: Empagliflozin (Matched to DPP-4) - South Korea vs DPP-4 (Matched to Empagliflozin) - South Korea; Outpatient healthcare visits - South Korea; Test type: Other; Rate Ratio = 0.97, 95% CI 2-sided [0.96 to 0.97] — Poisson regression model was used
Statistical Analysis 24: Comparison: Empagliflozin (Matched to DPP-4) - Norway vs DPP-4 (Matched to Empagliflozin) - Norway; Outpatient healthcare visits - Norway; Test type: Other; Rate Ratio = 0.96, 95% CI 2-sided [0.94 to 0.97]
Statistical Analysis 25: Comparison: Empagliflozin (Matched to DPP-4) - Spain vs DPP-4 (Matched to Empagliflozin) - Spain; Outpatient healthcare visit - Spain; Test type: Other; Rate Ratio = 0.88, 95% CI 2-sided [0.85 to 0.91] — Poisson regression model was used
Statistical Analysis 26: Comparison: Empagliflozin (Matched to DPP-4) - Sweden vs DPP-4 (Matched to Empagliflozin) - Sweden; Outpatient healthcare visits - Sweden; Test type: Other; Rate Ratio = 0.96, 95% CI 2-sided [0.94 to 0.98] — Poisson regression model was used
Statistical Analysis 27: Comparison: Empagliflozin (Matched to DPP-4) - Taiwan vs DPP-4 (Matched to Empagliflozin) - Taiwan; Outpatient healthcare visits - Taiwan; Test type: Other; Rate Ratio = 0.97, 95% CI 2-sided [0.94 to 1.00] — Poisson regression model was used

23. Secondary Outcome: Healthcare Resource Utilization (HCRU): Number of Any Prescription
Description: HCRU data were collected from seven of the 11 participating countries including Finland, Japan, South Korea, Norway, Spain, Sweden, and Taiwan. Outcomes captured as HCRU include pharmacy dispensations/prescriptions of different antidiabetic drugs, different drugs and prescriptions.
  HCRU outcomes were investigated for the matched cohort of empagliflozin/DPP-4 only. Due to possibly huge differences in healthcare systems and local practices, HCRU outcomes were presented descriptively by country as per prespecified analysis plan.
  For arms with 0 patients analyzed, no data was collected for the specific outcome in this country.
Time Frame: From index date until end of follow-up, up to 67 months.
Population: as for outcome 22
Measure: Number; unit: Prescription
Arm/Group | Empagliflozin (Matched to DPP-4) - Finland | DPP-4 (Matched to Empagliflozin) - Finland | Empagliflozin (Matched to DPP-4) - Japan | DPP-4 (Matched to Empagliflozin) - Japan | Empagliflozin (Matched to DPP-4) - South Korea | DPP-4 (Matched to Empagliflozin) - South Korea | Empagliflozin (Matched to DPP-4) - Norway | DPP-4 (Matched to Empagliflozin) - Norway | Empagliflozin (Matched to DPP-4) - Spain | DPP-4 (Matched to Empagliflozin) - Spain | Empagliflozin (Matched to DPP-4) - Sweden | DPP-4 (Matched to Empagliflozin) - Sweden | Empagliflozin (Matched to DPP-4) - Taiwan | DPP-4 (Matched to Empagliflozin) - Taiwan
Number analyzed (Participants) | 11801 | 11801 | 5592 | 5592 | 9072 | 9072 | 6344 | 6344 | 5865 | 5865 | 15785 | 15785 | 14048 | 14048
Prescription
  Pharmacy dispensations/prescriptions based on different antidiabetic drugs: number analyzed (Participants) | 0 | 0 | 5592 | 5592 | 9072 | 9072 | 0 | 0 | 0 | 0 | 0 | 0 | 14048 | 14048
  Pharmacy dispensations/prescriptions based on different antidiabetic drugs |  |  | 11243 | 11003 | 1417 | 1639 |  |  |  |  |  |  | 32341 | 29211
  Pharmacy dispensations/prescriptions based on different drugs: number analyzed (Participants) | 11801 | 11801 | 5592 | 5592 | 9072 | 9072 | 6344 | 6344 | 0 | 0 | 15785 | 15785 | 14048 | 14048
  Pharmacy dispensations/prescriptions based on different drugs | 80691 | 96770 | 64297 | 72589 | 113596 | 114278 | 53909 | 60072 |  |  | 125423 | 151096 | 188340 | 187291
  Pharmacy dispensations/prescriptions based on prescriptions | 259400 | 341506 | 41979 | 46888 | 93395 | 93602 | 174824 | 235661 | 37679 | 40448 | 430360 | 653294 | 207455 | 208526
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4) - Japan vs DPP-4 (Matched to Empagliflozin) - Japan; Pharmacy dispensations/prescriptions based on different antidiabetic drugs - Japan; Test type: Other; Rate Ratio = 0.91, 95% CI 2-sided [0.89 to 0.94] — Poisson regression model was used
Statistical Analysis 2: Comparison: Empagliflozin (Matched to DPP-4) - South Korea vs DPP-4 (Matched to Empagliflozin) - South Korea; Pharmacy dispensations/prescriptions based on different antidiabetic drugs - South Korea; Test type: Other; Rate Ratio = 0.86, 95% CI 2-sided [0.81 to 0.93] — Poisson regression model was used
Statistical Analysis 3: Comparison: Empagliflozin (Matched to DPP-4) - Taiwan vs DPP-4 (Matched to Empagliflozin) - Taiwan; Pharmacy dispensations/prescriptions based on different antidiabetic drugs - Taiwan; Test type: Other; Rate Ratio = 1.09, 95% CI 2-sided [1.08 to 1.11] — Poisson regression model was used
Statistical Analysis 4: Comparison: Empagliflozin (Matched to DPP-4) - Finland vs DPP-4 (Matched to Empagliflozin) - Finland; Pharmacy dispensations/prescriptions based on different drugs - Finland; Test type: Other; Rate Ratio = 1.11, 95% CI 2-sided [1.10 to 1.12] — Poisson regression model was used
Statistical Analysis 5: Comparison: Empagliflozin (Matched to DPP-4) - Japan vs DPP-4 (Matched to Empagliflozin) - Japan; Pharmacy dispensations/prescriptions based on different drugs - Japan; Test type: Other; Rate Ratio = 0.82, 95% CI 2-sided [0.81 to 0.83] — Poisson regression model was used
Statistical Analysis 6: Comparison: Empagliflozin (Matched to DPP-4) - South Korea vs DPP-4 (Matched to Empagliflozin) - South Korea; Pharmacy dispensations/prescriptions based on different drugs - South Korea; Test type: Other; Rate Ratio = 0.99, 95% CI 2-sided [0.99 to 1.00] — Poisson regression model was used
Statistical Analysis 7: Comparison: Empagliflozin (Matched to DPP-4) - Norway vs DPP-4 (Matched to Empagliflozin) - Norway; Pharmacy dispensations/prescriptions based on different drugs - Norway; Test type: Other; Rate Ratio = 1.12, 95% CI 2-sided [1.11 to 1.14] — Poisson regression model was used
Statistical Analysis 8: Comparison: Empagliflozin (Matched to DPP-4) - Sweden vs DPP-4 (Matched to Empagliflozin) - Sweden; Pharmacy dispensations/prescriptions based on different drugs - Sweden; Test type: Other; Rate Ratio = 1.26, 95% CI 2-sided [1.25 to 1.27] — Poisson regression model was used
Statistical Analysis 9: Comparison: Empagliflozin (Matched to DPP-4) - Taiwan vs DPP-4 (Matched to Empagliflozin) - Taiwan; Pharmacy dispensations/prescriptions based on different drugs - Taiwan; Test type: Other; Rate Ratio = 1.00, 95% CI 2-sided [0.98 to 1.02] — Poisson regression model was used
Statistical Analysis 10: Comparison: Empagliflozin (Matched to DPP-4) - Finland vs DPP-4 (Matched to Empagliflozin) - Finland; Pharmacy dispensations/prescriptions based on prescriptions - Finland; Test type: Other; Rate Ratio = 1.01, 95% CI 2-sided [1.01 to 1.02] — Poisson regression model was used
Statistical Analysis 11: Comparison: Empagliflozin (Matched to DPP-4) - Japan vs DPP-4 (Matched to Empagliflozin) - Japan; Pharmacy dispensations/prescriptions based on prescriptions - Japan; Test type: Other; Rate Ratio = 0.83, 95% CI 2-sided [0.82 to 0.84] — Poisson regression model was used
Statistical Analysis 12: Comparison: Empagliflozin (Matched to DPP-4) - South Korea vs DPP-4 (Matched to Empagliflozin) - South Korea; Pharmacy dispensations/prescriptions based on prescriptions - South Korea; Test type: Other; Rate Ratio = 1.00, 95% CI 2-sided [0.99 to 1.01] — Poisson regression model was used
Statistical Analysis 13: Comparison: Empagliflozin (Matched to DPP-4) - Norway vs DPP-4 (Matched to Empagliflozin) - Norway; Pharmacy dispensations/prescriptions based on prescriptions - Norway; Test type: Other; Rate Ratio = 0.93, 95% CI 2-sided [0.92 to 0.93] — Poisson regression model was used
Statistical Analysis 14: Comparison: Empagliflozin (Matched to DPP-4) - Spain vs DPP-4 (Matched to Empagliflozin) - Spain; Pharmacy dispensations/prescriptions based on prescriptions - Spain; Test type: Other; Rate Ratio = 0.86, 95% CI 2-sided [0.84 to 0.87] — Poisson regression model was used
Statistical Analysis 15: Comparison: Empagliflozin (Matched to DPP-4) - Sweden vs DPP-4 (Matched to Empagliflozin) - Sweden; Pharmacy dispensations/prescriptions based on prescriptions - Sweden; Test type: Other; Rate Ratio = 1.00, 95% CI 2-sided [1.00 to 1.00] — Poisson regression model was used

24. Secondary Outcome: Total Healthcare Costs - Finland, Norway, Sweden
Description: Total healthcare cost include costs for emergency room visits, first inpatient stay, all-cause hospital admissions, outpatient healthcare visits and pharmacy dispensations/prescriptions of different antidiabetic drugs, different drugs and prescriptions. Total healthcare costs for Finland, Norway and Sweden are reported in Euro per year.
  Due to possible huge differences in healthcare systems, cost of care outcomes are presented by country as prespecified in the analysis plan.
Time Frame: From index date until end of follow-up, up to 67 months.
Population: Only patients who were included in the matched cohort of empagliflozin/DPP-4i from Finland, Norway and Sweden. Cost are presented descriptively by country as per prespecified analysis plan.
Measure: Median (Inter-Quartile Range); unit: Euro per year
Arm/Group | Empagliflozin (Matched to DPP-4) - Finland | DPP-4 (Matched to Empagliflozin) - Finland | Empagliflozin (Matched to DPP-4) - Norway | DPP-4 (Matched to Empagliflozin) - Norway | Empagliflozin (Matched to DPP-4) - Sweden | DPP-4 (Matched to Empagliflozin) - Sweden
Number analyzed (Participants) | 11801 | 11801 | 6344 | 6344 | 15785 | 15785
Euro per year | 857 [270.2 to 2468.3] | 1356 [467.9 to 3677.8] | 1058 [452.8 to 2689.2] | 1336 [547.4 to 3678] | 658 [225.4 to 1771.9] | 1036 [418.3 to 2787.8]
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4) - Finland vs DPP-4 (Matched to Empagliflozin) - Finland; Total cost - Finland; Test type: Other; Rate Ratio = 0.89, 95% CI 2-sided [0.83 to 0.94] — Poisson regression model was used
Statistical Analysis 2: Comparison: Empagliflozin (Matched to DPP-4) - Norway vs DPP-4 (Matched to Empagliflozin) - Norway; Total costs - Norway; Test type: Other; Rate Ratio = 0.98, 95% CI 2-sided [0.86 to 1.12] — Poisson regression model was used
Statistical Analysis 3: Comparison: Empagliflozin (Matched to DPP-4) - Sweden vs DPP-4 (Matched to Empagliflozin) - Sweden; Total costs - Sweden; Test type: Other; Rate Ratio = 0.98, 95% CI 2-sided [0.92 to 1.05] — Poisson regression model was used

25. Secondary Outcome: Total Healthcare Cost - Japan
Description: Total healthcare costs include costs for emergency room visits, first inpatient stay, all-cause hospital admissions, outpatient healthcare visits and pharmacy dispensations/prescriptions of different antidiabetic drugs, different drugs and prescriptions.
  Total healthcare cost for Japan are reported in Japanese Yen (JPY) per year.
  Due to possible huge differences in healthcare systems, cost of care outcomes are presented by country as prespecified in the analysis plan.
Time Frame: From index date until end of follow-up, up to 67 months.
Population: Only patients who were included in the matched cohort of empagliflozin/DPP-4i from Japan. Costs are presented descriptively by country as per prespecified analysis plan.
Measure: Median (Inter-Quartile Range); unit: JPY per year
Arm/Group | Empagliflozin (Matched to DPP-4) - Japan | DPP-4 (Matched to Empagliflozin) - Japan
Number analyzed (Participants) | 5592 | 5592
JPY per year | 91867 [15329.9 to 320776] | 63773 [9773.9 to 260629.4]
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4) - Japan vs DPP-4 (Matched to Empagliflozin) - Japan; Test type: Other; Rate Ratio = 0.84, 95% CI 2-sided [0.80 to 0.88] — Poisson regression model was used

26. Secondary Outcome: Total Healthcare Cost - South Korea
Description: Total healthcare costs include costs for emergency room visits, first inpatient stay, all-cause hospital admissions, outpatient healthcare visits and pharmacy dispensations/prescriptions of different antidiabetic drugs, different drugs and prescriptions.
  Total healthcare costs for South Korea are reported in 1000 Korean Won (KRW) per year.
  Due to possible huge differences in healthcare systems, cost of care outcomes are presented by country as prespecified in the analysis plan.
Time Frame: From index date until end of follow-up, up to 67 months.
Population: Only patients who were included in the matched cohort of empagliflozin/DPP-4i from South Korea. Cost are presented descriptively by country as per prespecified analysis plan.
Measure: Median (Inter-Quartile Range); unit: 1000 KRW per year
Arm/Group | Empagliflozin (Matched to DPP-4) - South Korea | DPP-4 (Matched to Empagliflozin) - South Korea
Number analyzed (Participants) | 9072 | 9072
1000 KRW per year | 214 [58.15 to 557.23] | 220 [58.62 to 636.53]
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4) - South Korea vs DPP-4 (Matched to Empagliflozin) - South Korea; Total costs - South Korea; Test type: Other; Rate Ratio = 0.76, 95% CI 2-sided [0.34 to 1.68] — Poisson regression model was used

27. Secondary Outcome: Total Healthcare Cost - Taiwan
Description: Total healthcare costs include costs for emergency room visits, first inpatient stay, all-cause hospital admissions, outpatient healthcare visits and pharmacy dispensations/prescriptions of different antidiabetic drugs, different drugs and prescriptions.
  Total healthcare cost for Taiwan are reported in United States Dollar (USD) per year.
  Due to possible huge differences in healthcare systems, cost of care outcomes are presented by country as prespecified in the analysis plan.
Time Frame: From index date until end of follow-up, up to 67 months.
Population: Only patients who were included in the matched cohort of empagliflozin/DPP-4i from Taiwan. Costs are presented descriptively by country as per prespecified analysis plan.
Measure: Median (Inter-Quartile Range); unit: USD per year
Arm/Group | Empagliflozin (Matched to DPP-4) - Taiwan | DPP-4 (Matched to Empagliflozin) - Taiwan
Number analyzed (Participants) | 14048 | 14048
USD per year | 530 [157.9 to 1330.1] | 431 [120.6 to 1205.6]
Statistical Analysis 1: Comparison: Empagliflozin (Matched to DPP-4) - Taiwan vs DPP-4 (Matched to Empagliflozin) - Taiwan; Total costs - Taiwan; Test type: Other; Rate Ratio = 0.97, 95% CI 2-sided [0.92 to 1.03] — Poisson regression model was used

ADVERSE EVENTS:
Time Frame: Not applicable for serious and other adverse events. [All-cause mortality]: Up to 86 months.
Description: This is a non-interventional study using secondary data. Serious and other adverse events were not planned to be collected and reported. The "0" in Serious and Other Adverse Events sections refers to "not applicable".
  [All-cause mortality]: All patients included in the study, who were either new user of any SGLT-2i (incl. empagliflozin) or DPP-4i. Deaths are reported by SGLT-2i (incl. empagliflozin) and DPP-4i group, as specified in statistical analysis plan.
Arm/Group | SGLT-2i (Incl. Empa) (Matched to DPP-4i) | DPP-4i (Matched to SGLT-2i)
All-Cause Mortality (participants affected / at risk) | 1371/163812 | 2524/163812
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT03817463/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT03817463/SAP_001.pdf